CLINICAL TRIAL: NCT07319052
Title: Effects of β-Alanine Supplementation on Kickboxing-Specific Anaerobic Performance, Neuromuscular Power, and Strength Endurance: A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: β-Alanine for Kickboxing Anaerobic Performance
Acronym: BA-KAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Salih ÇABUK (Other)
Responsible Party: Sponsor-Investigator, Salih ÇABUK, Research Assistant, Erzurum Technical University
Organization: Erzurum Technical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ETU-BETAALANINE-2025; 06/5/21.04.2025 (Other: Erzurum Technical University)
Record Dates: First submitted 2025-12-21; First posted 2026-01-06 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Athletic Performance Enhancement (Kickboxing); Anaerobic Performance; Strength Endurance; Neuromuscular Power; Nutritional Supplementation (β-Alanine)
Keywords: β-alanine; Kickboxing Anaerobic Speed Test; KAST; randomized double-blind placebo-controlled
MeSH Terms: interventions — Flour

STUDY DESIGN:
Intervention Model Description: Participants are randomized 1:1 (stratified by competitive level) to β-alanine or placebo in a parallel-group design. Allocation is concealed with blocked randomization; participants, investigators, coaches, and outcome assessors are blinded. No crossover or clustering; outcomes are assessed at baseline and after 4 weeks of supplementation.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Both participants and investigators are blinded to group allocation. Supplements are pre-packaged in identical, coded containers prepared by an independent staff member not involved in testing or data analysis. Coaches supervising the training sessions and all outcome assessors analyzing video and performance data are also blinded to the intervention codes until statistical analyses are complete.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- β-Alanine Supplementation (Experimental): Participants receive 6.4 g of β-alanine per day for 4 weeks (e.g., 4 × 1.6 g divided doses). The supplement is provided as Hardline β-Alanine (Hardline Nutrition, Türkiye), standardized for active ingredient content.
  Interventions: Dietary Supplement: β-Alanine
- Rice Flour (Placebo Comparator): Participants receive a visually identical, flavor-matched placebo composed of rice flour, dosed equivalently to the experimental group (6.4 g·day-¹ for 4 weeks).
  Interventions: Dietary Supplement: Rice Flour (Placebo)

INTERVENTIONS:
Dietary Supplement: β-Alanine — Participants in the experimental group will receive 6.4 grams of β-alanine per day for 4 weeks, administered orally in four divided doses (1.6 g each). The supplement used is a commercially available β-alanine formulation (Hardline Nutrition, Türkiye), standardized for purity and active ingredient content. The dosing protocol follows established guidelines from prior ergogenic studies in athletes. Supplementation is supervised by the research team, and adherence is monitored weekly.
  Arms: β-Alanine Supplementation
Dietary Supplement: Rice Flour (Placebo) — Participants in the placebo group will receive 6.4 grams of rice flour per day for 4 weeks, divided into four equal doses (1.6 g each) and identical in appearance, packaging, and flavor to the β-alanine supplement. The placebo is prepared and coded by an independent staff member to maintain double-blind conditions. All participants consume their assigned supplement orally each day under the same schedule, maintaining their normal training and diet routines.
  Arms: Rice Flour

SUMMARY:
This randomized, double-blind, placebo-controlled parallel-group trial will evaluate whether four weeks of β-alanine (BA) supplementation improves sport-specific anaerobic performance, neuromuscular power, and strength endurance in trained male kickboxers. β-Alanine is the rate-limiting precursor for skeletal muscle carnosine, an intramuscular buffer that can attenuate exercise-induced acidosis during repeated high-intensity efforts. Because kickboxing involves brief, repeated striking sequences with high glycolytic demand, BA may represent a practical, legal ergogenic aid for this population.

Twenty-eight adult male kickboxers will be randomized (stratified) to BA (6.4 g·day-¹) or placebo for 4 weeks while maintaining habitual training and diet. Assessments will occur at baseline and post-intervention under standardized laboratory conditions and time-of-day control. The primary outcome is the total time on the Kickboxing Anaerobic Speed Test (KASTtotal; five consecutive sets of a validated four-technique striking combination with 10-s passive recovery). Secondary outcomes include best single-set time (KASTbest), individual set times (KAST₁-₅), Performance Decrement Index (PDI), countermovement jump (CMJ) and squat jump (SJ) height, and upper-body strength endurance (maximal push-ups and pull-ups performed to strict standards). Timing is determined from 25-fps video with frame-level analysis; jump height is derived via a validated smartphone application.

Adverse events-particularly transient paresthesia-will be monitored throughout. The main analysis will use two-way repeated-measures ANOVA (group × time) with partial eta-squared to quantify effects; assumption checks and correction procedures will be applied as appropriate. BA will yield greater improvements than placebo in KASTtotal and upper-body strength endurance, with limited changes expected for jump performance.

DETAILED DESCRIPTION:
Rationale and Background: β-Alanine supplementation increases intramuscular carnosine, enhancing intracellular buffering capacity and potentially preserving excitation-contraction coupling during high-intensity, repeated efforts. Kickboxing competition is characterized by short striking bouts, rapid direction changes, and high glycolytic contribution-conditions under which increased buffering may translate to meaningful performance benefits. Prior work in combat sports has reported ergogenic effects of BA; however, evidence in kickboxing using a validated sport-specific test remains limited. This trial addresses that gap using the Kickboxing Anaerobic Speed Test (KAST), which offers strong ecological validity for combat athletes.

Design and Setting: Randomized, double-blind, placebo-controlled, parallel-group clinical trial with two assessment time points (pre, post). Participants continue usual training under coach supervision and are instructed to avoid other ergogenic aids and caffeine for 24 h before testing. All testing is performed under standardized environmental conditions (temperature and humidity controlled) and at the same time of day (±1 h) to minimize circadian and residual fatigue effects.

Participants: Twenty-eight healthy adult male kickboxers with ≥5 years of systematic training and active competition in the prior year. Key exclusions include musculoskeletal injury limiting high-intensity exercise, cardiometabolic or respiratory disease, β-alanine intolerance, and recent use of overlapping supplements. Written informed consent is obtained. The protocol complies with the Declaration of Helsinki and local ethics approval.

Interventions Experimental: β-alanine, 6.4 g·day-¹ for 4 weeks (e.g., divided doses). Comparator: Appearance-matched placebo (rice flour), same schedule. Products are dispensed in coded containers to preserve blinding of participants, investigators, and outcome assessors.

Outcome Measures Primary: KASTtotal (s), computed as the sum of five consecutive sets of a standardized four-technique combination performed at maximal effort with 10-s passive recovery. Timing starts at first bag contact and ends after the final kick; performance is video-recorded at 25 fps and analyzed frame-by-frame.

Secondary: KASTbest (best of two maximal sets separated by 5-min recovery), individual set times KAST₁-₅, PDI (%) = KASTtotal/(KASTbest × 5) × 100, CMJ and SJ height (hands on hips; validated smartphone app), and maximal push-ups and pull-ups (strict form criteria). Adverse events and tolerability-especially paresthesia-are recorded throughout.

Procedures and Standardization: A familiarization session precedes baseline testing. Warm-up includes light aerobic activity, dynamic drills, plyometrics, mobility work, and shadowboxing following a scripted sequence. Standardized verbal encouragement and rest intervals are used. Technique order for KAST is fixed; any deviation leads to trial termination and repeat after enforced rest.

Sample Size and Statistical Analysis: An a priori power analysis for a medium within-between interaction (α=0.05, power 0.80) indicated a minimum sample of 24; the target enrollment of 28 provides adequate sensitivity. Baseline between-group differences are assessed by independent t-tests (effect size: Hedges' g). The primary inferential model is a two-way repeated-measures ANOVA (group × time) for each outcome, reporting F(1,26), p values, and partial eta-squared (ηp²) with conventional magnitude thresholds. Assumptions are tested (Shapiro-Wilk, Levene, Mauchly); Greenhouse-Geisser corrections are applied as needed. When interactions are significant, simple-effects tests with Bonferroni adjustment localize differences.

Safety and Monitoring: This is a low-risk nutrition study in trained athletes. The most common expected adverse effect is transient paresthesia, which will be monitored via spontaneous reports and direct questioning. Any unexpected or serious events will be evaluated and reported per institutional policy; supplementation may be paused or discontinued at investigator discretion.

Expected Impact and Limitations: BA to reduce KASTtotal and improve push-up and pull-up performance versus placebo, with minimal changes in CMJ/SJ. Limitations include the absence of direct physiological verification of carnosine accrual (e.g., muscle biopsy) and lack of concurrent lactate or pH measures, which constrain mechanistic inference. Nonetheless, by deploying a validated, sport-specific performance test with rigorous control of confounders and blinded assessment, this trial aims to provide clinically relevant, ecologically valid evidence for practitioners working with combat sport athletes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male kickboxers aged 18-35 years
* Minimum 5 years of systematic kickboxing training experience
* Actively engaged in competition or structured training within the last 12 months
* Free from any musculoskeletal injuries, metabolic, cardiovascular, or respiratory disorders that could affect high-intensity exercise performance
* Not currently taking any ergogenic aids, nutritional supplements, or medications known to influence performance or recovery
* Willing to maintain habitual diet and training routines throughout the study period
* Provided written informed consent before participation

Exclusion Criteria:

* Current or recent (<6 months) musculoskeletal injury preventing maximal effort performance
* Metabolic, cardiovascular, or respiratory conditions that may increase risk during high-intensity activity
* Known allergy or intolerance to β-alanine
* Use of performance-enhancing supplements (e.g., creatine, caffeine, sodium bicarbonate, beta-alanine) in the past 4 weeks
* Any neurological, psychiatric, or endocrine disorder affecting physical performance or adherence
* Inability or unwillingness to comply with supplementation protocol or testing procedures

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2025-04-30 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-06-04 (Actual)

PRIMARY OUTCOMES:
Total Time on Kickboxing Anaerobic Speed Test (KASTtotal) | Baseline (Pre-supplementation) and after 4 weeks of supplementation (Post-intervention).
  KASTtotal represents the cumulative time (in seconds) required to complete five consecutive sets of a standardized four-technique striking combination (jab-roundhouse-cross-roundhouse) performed at maximal intensity, with 10 seconds of passive recovery between sets. Timing begins at the first strike and ends at the completion of the final kick. This outcome reflects total anaerobic performance capacity under repeated high-intensity conditions specific to kickboxing.

SECONDARY OUTCOMES:
Best Single-Set Time (KASTbest) | Baseline and Week 4
  Fastest time achieved across two maximal-effort sets of the KAST protocol, separated by 5 minutes of rest.
Countermovement Jump Height (CMJ) | Baseline and Week 4
  Vertical jump height (cm) measured using the validated MyJump2 mobile application based on flight time, with hands on hips. Reflects lower-limb explosive power.
Squat Jump Height (SJ) | Baseline and Week 4
  Vertical jump height (cm) measured from a static 90° knee flexion position held for 3 seconds prior to the jump, assessed using MyJump2.
Push-up Repetitions | Baseline and Week 4
  Maximum number of continuous, correctly performed push-ups maintaining full elbow extension and rigid body alignment.
Pull-up Repetitions | Baseline and Week 4
  Maximum number of continuous pull-ups performed with pronated grip, full arm extension at the start, and chin passing the bar at the top.

CONTACTS AND LOCATIONS:
Locations (1):
- Erzurum Technical University, Sport Laboratory, Erzurum, Yakutiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data (IPD) will not be shared publicly, as this study involves a relatively small sample of competitive athletes whose anonymized data could still be indirectly identifiable due to performance metrics and demographic characteristics. Only aggregated and de-identified summary results will be reported in peer-reviewed publications and conference presentations. Upon reasonable request, group-level statistical data or analysis code may be shared with qualified researchers following institutional and ethical approval procedures.